CLINICAL TRIAL: NCT02419313
Title: Investigation of the Efficacy and Safety of IncobotulinumtoxinA (Xeomin) in Parkinson's Disease Tremor: A Customized Approach
Brief Title: Investigation of the Efficacy and Safety of IncobotulinumtoxinA (Xeomin) in Parkinson's Tremor: A Customized Approach
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1206010370
Record Dates: First submitted 2014-01-27; First posted 2015-04-17 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Parkinson; Tremor
Keywords: Tremor; Parkinson; botulinum; Xeomin
MeSH Terms: conditions — Tremor | interventions — incobotulinumtoxinA; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo, then Xeomin (Active Comparator): Subjects randomized to receive the placebo ( saline) will receive an equivalent volume as the active study drug (1cc). The injections will be into -10 hand and forearm muscles. A series of rating scale and an examination will take place prior to treatment and at 4 and 8 weeks post treatment. The subject will then cross over to an Active Intervention arm to receive incobotulinumtoxinA which will be injected in the same pattern as the saline.
  Interventions: Drug: incobotulinumtoxinA; Drug: Saline
- Xeomin, then Placebo (Active Comparator): Subjects will all receive injections with incobotulinumtoxinA injections, 100unit/cc into 6-10 muscles of the forearm. A series of rating scale and an examination will take place prior to treatment and at 4 and 8 weeks post treatment. These subjects will then cross over and receive placebo ( saline) in the same distribution as their second treatment.
  Interventions: Drug: incobotulinumtoxinA; Drug: Saline

INTERVENTIONS:
Drug: incobotulinumtoxinA — Subjects randomized to the active drug intervention arm will receive incobotulinumtoxinA (Xeomin). A series of rating scales and examinations will take place prior to treatment and for 24 weeks after treatment. At 12 weeks the subjects will cross over to the placebo (saline) arm.
  Other Names: Xeomin
Drug: Saline — same volume as injected for incobotulinum toxin A into forearm muscles under EMG guidance.
  Other Names: Placebo

SUMMARY:
The scientific aim of this study is to investigate the efficacy and safety of incobotulinumtoxinA (Xeomin-Merz Pharmaceuticals) in the tremor of Parkinson"s disease. Our hypothesis is that injection of Xeomin into the muscles of arm, forearm and hand decreases the tremor amplitude and frequency leading to improvement of the patient"s function.

DETAILED DESCRIPTION:
This is an investigator initiated, randomized, double blind, placebo controlled, cross over study which is supported by Merz pharmaceuticals. Patients with Parkinson"s disease (at Yale Neurology and Movement disorders clinics) will be approached by the members of the research team (PI and sub-investigators) to see if they meet inclusion and exclusion criteria and wish to participate in the study.

If eligible and consented to participate in the study, there will be a series of questionaires, examinations and treatment sessions.

ELIGIBILITY:
Inclusion Criteria.

1. Age more than 18 years
2. Both sexes
3. all races/ethnic groups.
4. Meeting the clinical diagnosis of Parkinson's disease with presence of moderate to severe Parkinson tremor that is refractory to standard medical treatments and which limits the patient"s functionality and/or poses significant discomfort.
5. Subjects who are able to read, speak, and understand English.

Exclusion Criteria.

1. Existing significant acute medical condition (i.e. cardiovascular, endocrine, hematologic, neoplastic, infectious, or autoimmune disorders) or significant swallowing or breathing difficulties.
2. Pregnancy or planned pregnancy (determined by urine pregnancy test).
3. Active breast feeding.
4. Enrollment in any clinical trial (currently or within the past 3 months) in which treatments are imposed by a protocol.
5. Any subject for whom botulinum toxin treatment would be contraindicated; known allergy or sensitivity to medication.
6. Subjects who are younger than 18 years of age. Neuromuscular-junction disorders.
7. Evidence of acute pathology in neuro-imaging.
8. Axis I diagnosis determined by a neurologist or psychiatrist.
9. Use of Anesthetic medications within two weeks and corticosteroid injections within 4 weeks of enrollment.
10. Those who received botulinum toxin injections in the past 4 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bahman Jabbari, MD, Principal Investigator — Yale University
Locations (1):
- Yale Neurology, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mittal SO, Machado D, Richardson D, Dubey D, Jabbari B. Botulinum Toxin in Parkinson Disease Tremor: A Randomized, Double-Blind, Placebo-Controlled Study With a Customized Injection Approach. Mayo Clin Proc. 2017 Sep;92(9):1359-1367. doi: 10.1016/j.mayocp.2017.06.010. Epub 2017 Aug 5. PMID 28789780

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First, Then Incobotulinumtoxin A: Subjects will all receive injections with saline first. At 12 weeks, these subjects will then cross over and receive Xeomin in the same distribution as their second treatment.
- Incobotulinumtoxin A First, Then Placebo: Subjects will all receive injections with incobotulinumtoxinA injections first. At 12 weeks, these subjects will then cross over and receive placebo in the same distribution as their second treatment.
Period: First Intervention
Arm/Group | Placebo First, Then Incobotulinumtoxin A | Incobotulinumtoxin A First, Then Placebo
Started | 18 | 15
Completed | 16 | 15
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Period: Second Intervention
Arm/Group | Placebo First, Then Incobotulinumtoxin A | Incobotulinumtoxin A First, Then Placebo
Started | 16 | 15
Completed | 15 | 15
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: double blind cross over study aimed at 30 patients 33 enrolled- 30 completed
Groups:
- All Study Participants: All participants included in this crossover design.
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 12
Age, Continuous [Mean (Full Range); unit: years] | 61.7 [52 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Unified Parkinsons Disease Rating Scale (UPDRS) Tremor Scale
Description: The primary outcome measure in this protocol is significant improvement of tremor (equal or over 2 grade improvement) of the Unified Parkinson's Disease Rating Scale 4 weeks after Xeomin injection. The score is 0 to 4 , ) being no tremor and 4 severe tremor. The higher the score, the more severe the tremor.
Time Frame: 4 weeks
Measure: Number; unit: participants
Groups:
- Placebo, Saline: Subjects randomized to receive the placebo ( saline) will receive an equivalent volume as the active study drug (1cc). The injections will be into -10 hand and forearm muscles. A series of rating scale and an examination will take place prior to treatment and at 4 and 8 weeks post treatment. The subject will then cross over to an Active Intervention arm to receive incobotulinumtoxinA which will be injected in the same pattern as the saline.
  Saline: same volume as injected for incobotulinum toxin A into forearm muscles under EMG guidance.
- incobotulinumtoxinA, Xeomin: Subjects will all receive injections with incobotulinumtoxinA injections, 100unit/cc into 6-10 muscles of the forearm. A series of rating scale and an examination will take place prior to treatment and at 4 and 8 weeks post treatment. These subjects will then cross over and receive placebo ( saline) in the same distribution as their second treatment.
  incobotulinumtoxinA: Subjects randomized to the active drug intervention arm will receive incobotulinumtoxinA (Xeomin). A series of rating scales and examinations will take place prior to treatment and for 24 weeks after treatment. At 12 weeks the subjects will cross over to the placebo (saline) arm.
Arm/Group | Placebo, Saline | incobotulinumtoxinA, Xeomin
Number analyzed (Participants) | 30 | 30
participants | 0 | 8
Statistical Analysis 1: Comparison: Placebo, Saline vs incobotulinumtoxinA, Xeomin; Test type: Superiority or Other; p = 0.0007, Fisher Exact

2. Secondary Outcome: Number of Patients Whose Patient Global Impression of Change (PGIC) Improved
Description: The PGIC is a 7 point scale that requires the clinician to assess how much the patient's pain has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as:
  No change (or condition has gotten worse) (1) Almost the same, hardly any change at all (2) A little better, but no noticeable change (3) Somewhat better, but the change has not made any real difference (4) Moderately better, and a slight but noticeable change (5) Better and a definite improvement that has made a real and worthwhile difference (6) A great deal better and a considerable improvement that has made all the difference (7)improved
  This outcome is number of patients who chose a 6 or above on the PGIC 6 weeks after treatment.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Placebo, Saline | incobotulinumtoxinA, Xeomin
Number analyzed (Participants) | 30 | 30
participants | 0 | 10
Statistical Analysis 1: Comparison: Placebo, Saline vs incobotulinumtoxinA, Xeomin; Test type: Superiority or Other; p = 0.0008, Fisher Exact

3. Secondary Outcome: Patients With Significant Improvement in Unified Parkinsons Disease Rating Tremor Scale
Description: This scale measures the amplitude of the tremor. For instance tremor of more than 4cm oscillation is grade 4. UPDRS tremor scale is 0-4 , 4 being severe tremor. Significant improvement for this protocol considered two grades of improvement .
Time Frame: 4 Weeks
Measure: Number; unit: participants
Arm/Group | Placebo, Saline | incobotulinumtoxinA, Xeomin
Number analyzed (Participants) | 30 | 30
participants | 0 | 8
Statistical Analysis 1: Comparison: Placebo, Saline vs incobotulinumtoxinA, Xeomin; Test type: Superiority or Other; p = 0.0105, Fisher Exact

ADVERSE EVENTS:
Time Frame: 6 months Every 4 weeks regular check up Patient to call immediately if adverse effect happened
Description: as above
Arm/Group | Placebo, Saline | incobotulinumtoxinA, Xeomin
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 3/33 | 3/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo, Saline (N=33) | incobotulinumtoxinA, Xeomin (N=33)
muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No